CLINICAL TRIAL: NCT00797303
Title: The Effect of Bevacizumab on Corneal Neovascularization
Acronym: BQ-1-08-ARVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, Clinical Professor, Instituto de Olhos de Goiania
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BQ-1-08-ARVO
Record Dates: First submitted 2008-11-22; First posted 2008-11-25 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Corneal Neovascularization
Keywords: bevacizumab; cornea; neovascularization
MeSH Terms: conditions — Corneal Neovascularization; Corneal Diseases; Neovascularization, Pathologic | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): A single intraoperative subconjunctival application of bevacizumab and 2 months follow-up
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — subconjunctival injection of 1.25 mg bevacizumab and had a follow-up of at least 2 months

SUMMARY:
Eight patients with corneal neovascularization were treated with subconjunctival injection of 1.25 mg bevacizumab and had a follow-up of at least 2 months. All patients had persistent corneal neovascularization for at least 6 months unresponsive to other treatments. Patients were monitored by ophthalmic exam and anterior segment photography.

DETAILED DESCRIPTION:
To evaluate the effect of repeated subconjunctival bevacizumab (Avastin®, Roche, Rio de Janeiro, Brazil) on inflammatory corneal neovascularization.

Eight patients with corneal neovascularization were treated with subconjunctival injection of 1.25 mg bevacizumab and had a follow-up of at least 2 months. All patients had persistent corneal neovascularization for at least 6 months unresponsive to other treatments. Patients were monitored by ophthalmic exam and anterior segment photography.

ELIGIBILITY:
Inclusion Criteria:

* Corneal Neovascularization
* Stable lesion

Exclusion Criteria:

* Diabetes
* Autoimmune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The Effect of Bevacizumab on Corneal Neovascularization | Compare the results
  Eight patients with corneal neovascularization were treated with subconjunctival injection of 1.25 mg bevacizumab and had a follow-up of at least 2 months. All patients had persistent corneal neovascularization for at least 6 months unresponsive to other treatments. Patients were monitored by ophthalmic exam and anterior segment photography

CONTACTS AND LOCATIONS:
Overall Officials: Belquiz A Nassaralla, PhD, Study Chair — Instituto de Olhos de Goiânia